CLINICAL TRIAL: NCT02662413
Title: To Determine the Measurement Properties of the ACT in an Adolescent Population With Persistent Asthma Followed at a Subspecialty Clinic.
Brief Title: To Determine the Validity of the ACT in an Adolescent Population With Persistent Asthma
Acronym: ACT2
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Academy of Allergy, Asthma, and Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: 15-1804
Record Dates: First submitted 2016-01-05; First posted 2016-01-25 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Validation of Asthma Control Questionnaire — This is an observational study so there is no planned intervention.

SUMMARY:
To determine the measurement profiles of the asthma control test (ACT) in an adolescent population with persistent asthma.

DETAILED DESCRIPTION:
Asthma is the most common chronic illness of childhood, and adolescents represent a group that is typically difficult to engage in self-management strategies. Adolescent asthmatics tend to have poor perception of symptoms and experience a higher rate of asthma deaths compared to younger children. Studies have shown that perceived severity of asthma symptoms is related to self-management in adolescents, who were less likely to receive appropriate treatment for asthma exacerbation's. This poor perception of asthma control is likely one cause of the disproportionate asthma mortality rates seen in adolescent patients.

Because asthma control is now the focus of asthma care, assessment of control is the critical step in appropriate management. The two domains of asthma control, impairment and risk, evaluate the role asthma plays in a patient's quality of life and functional capacity on an ongoing basis and the risk their asthma presents for future adverse events. Although the National Asthma Education and Prevention Program guidelines contain a rubric for asthma control based on these domains, thus representing the "gold standard" for asthma care, their utilization may be time-consuming and cumbersome to implement in primary care offices, and primary care providers may be unfamiliar with their use. For primary care practices following adolescent patients, it remains imperative that the tools being used to gauge asthma control be evaluated and validated in this at-risk population.

At this time, there are approximately 17 questionnaires available for use in the assessment of asthma control, although most are not well validated. Of these, the most widely validated and most commonly used instrument is the Asthma Control Test (ACT). The ACT is a self-administered questionnaire intended to assess the impairment domain over the past four weeks and is completed by patients starting at age 12 years. The ACT has five questions with an overall best score of 25. For primarily adult Caucasian populations, the ACT has been found to be a valid, reliable, and responsive instrument of asthma control, and cut-offs for controlled and not well controlled asthma (< 19) as well as minimal clinically important (MIC) differences (3 points) have been identified. The measurement properties of validity, reliability, and responsiveness are critical to the usefulness of any questionnaire in both clinical and research settings. However, measurement properties of the ACT are lacking in the adolescent asthma population.The landmark validation study for the ACT by Schatz et al was comprised of a large sample size of over 300 patients that showed that a cut-off score of 19 as distinguishing well-controlled versus not well-controlled asthmatics. However, the mean age was 35 for that study population, and concerns have been raised as to whether this cut-off is appropriate for adolescents in general. Recent studies examining use of the ACT in Caucasian and Hispanic adolescent populations have found higher optimal cut points to distinguish control classifications.

Lung function measures are included in the rubric of assessing asthma control by the NAEPP (National Asthma Education and Prevention Program). Per these recommendations, spirometry should be available to physicians caring for asthma patients and used with initiation of treatment, change in asthma control, and every one to two years. While sub-specialists often have access to spirometry, office-based spirometry is time-consuming, requires technical ability and staff training, equipment maintenance and calibration, and is not always available or feasible for use in primary care physician offices. Because spirometry may be of limited accessibility to primary care providers, questionnaires are quickly taking a leading role in asthma management. Studies of adolescent asthmatics reveal poor perception of asthma control leading to under-reporting of asthma symptoms and thus under-treatment of exacerbation's. This type of under-reporting reflects a false level of asthma control when queried by the ACT and leads to inappropriate medical management when spirometry is not utilized.

As exploratory endpoints, we will obtain fractional exhaled nitric oxide (FeNO) measurements shortly after spirometry is performed. Elevated FeNO indicates eosinophilic airway inflammation and assists in assigning the correct asthma phenotype, which can have implications for asthma management. We will also obtain nasal epithelial lining fluid (ELF) for collection of nasal cytokines and chemokines. This information is useful for expanding our current understanding of the inflammatory mediators involved in asthma-associated airway inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of persistent asthma
* Current treatment with appropriate therapy for persistent asthma symptoms per the NHLBI guidelines including daily controller medication with at least low dose inhaled corticosteroids
* Must live within convenient driving distance of the North Carolina Children's Specialty Clinic in Raleigh North Carolina or the EPA Human Studies Facility on University of North Carolina Campus in Chapel Hill North Carolina.

Exclusion Criteria:

* Unable to perform spirometry
* Other medical history or underlying health problems that would preclude participation.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children ages 12-18 with a physician diagnosis of persistent asthma living in a defined geographical area
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08-10 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Cohen's kappa | Baseline visit
  To determine the agreement of the ACT score at the standard cutpoint of >19 with physician assessment of control using Cohen's kappa.

SECONDARY OUTCOMES:
Sensitivity of ACT Questionnaire | follow-up visit (six weeks)
  A receiver-operating curve will be used to determine the best ACT cutpoint for assessment of control in this population. A logistic regression model will be used with 'control by physician' as the dependent variable and 'ACT score' as the independent variable. The model will include adjustment for repeated measures (baseline and 6 week visit).
Specificity of ACT Questionnaire | follow-up visit (six weeks)
  A receiver-operating curve will be used to determine the best ACT cutpoint for assessment of control in this population. A logistic regression model will be used with 'control by physician' as the dependent variable and 'ACT score' as the independent variable. The model will include adjustment for repeated measures (baseline and 6 week visit).
Cohen's kappa | follow-up visit (six weeks)
  To determine the agreement of the ACT score at the standard cutpoint of >19 with physician assessment of control using Cohen's kappa.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Burbank, MD, Principal Investigator — Fellow; Michelle Hernandez, MD, Study Director — Assistant Professor
Locations (2):
- United States (2):
  - UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina
  - NC Children's Specialty Clinic, 4414 Lake Boone Trail, Suite 505, Raleigh, North Carolina

REFERENCES:
- [Background] Raherison C, Tunon-de-Lara JM, Vernejoux JM, Taytard A. Practical evaluation of asthma exacerbation self-management in children and adolescents. Respir Med. 2000 Nov;94(11):1047-52. doi: 10.1053/rmed.2000.0888. PMID 11127490
- [Background] Larsen GL. Asthma in children. N Engl J Med. 1992 Jun 4;326(23):1540-5. doi: 10.1056/NEJM199206043262306. PMID 1579137
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Background] Cloutier MM, Schatz M, Castro M, Clark N, Kelly HW, Mangione-Smith R, Sheller J, Sorkness C, Stoloff S, Gergen P. Asthma outcomes: composite scores of asthma control. J Allergy Clin Immunol. 2012 Mar;129(3 Suppl):S24-33. doi: 10.1016/j.jaci.2011.12.980. PMID 22386507
- [Background] Juniper EF, Gruffydd-Jones K, Ward S, Svensson K. Asthma Control Questionnaire in children: validation, measurement properties, interpretation. Eur Respir J. 2010 Dec;36(6):1410-6. doi: 10.1183/09031936.00117509. Epub 2010 Jun 7. PMID 20530041
- [Background] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Background] Korn S, Both J, Jung M, Hubner M, Taube C, Buhl R. Prospective evaluation of current asthma control using ACQ and ACT compared with GINA criteria. Ann Allergy Asthma Immunol. 2011 Dec;107(6):474-9. doi: 10.1016/j.anai.2011.09.001. Epub 2011 Oct 5. PMID 22123375
- [Background] Schatz M, Sorkness CA, Li JT, Marcus P, Murray JJ, Nathan RA, Kosinski M, Pendergraft TB, Jhingran P. Asthma Control Test: reliability, validity, and responsiveness in patients not previously followed by asthma specialists. J Allergy Clin Immunol. 2006 Mar;117(3):549-56. doi: 10.1016/j.jaci.2006.01.011. PMID 16522452
- [Background] Thomas M, Kay S, Pike J, Williams A, Rosenzweig JR, Hillyer EV, Price D. The Asthma Control Test (ACT) as a predictor of GINA guideline-defined asthma control: analysis of a multinational cross-sectional survey. Prim Care Respir J. 2009 Mar;18(1):41-9. doi: 10.4104/pcrj.2009.00010. PMID 19240948
- [Background] Leung TF, Ko FW, Sy HY, Wong E, Li CY, Yung E, Hui DS, Wong GW, Lai CK. Identifying uncontrolled asthma in young children: clinical scores or objective variables? J Asthma. 2009 Mar;46(2):130-5. doi: 10.1080/02770900802468533. PMID 19253117
- [Background] Koolen BB, Pijnenburg MW, Brackel HJ, Landstra AM, van den Berg NJ, Merkus PJ, Hop WC, Vaessen-Verberne AA. Comparing Global Initiative for Asthma (GINA) criteria with the Childhood Asthma Control Test (C-ACT) and Asthma Control Test (ACT). Eur Respir J. 2011 Sep;38(3):561-6. doi: 10.1183/09031936.00173710. Epub 2011 Mar 15. PMID 21406508
- [Background] Shi Y, Tatavoosian AV, Aledia AS, George SC, Galant SP. Cut points for Asthma Control Tests in Mexican children in Orange County, California. Ann Allergy Asthma Immunol. 2012 Aug;109(2):108-13. doi: 10.1016/j.anai.2012.06.002. Epub 2012 Jul 4. PMID 22840251
- [Derived] Burbank AJ, Todoric K, Steele P, Rosen J, Zhou H, Frye M, Loughlin CE, Ivins S, Mills K, Massey LD, Reeve BB, Hernandez ML. Age and African-American race impact the validity and reliability of the asthma control test in persistent asthmatics. Respir Res. 2018 Aug 15;19(1):152. doi: 10.1186/s12931-018-0858-0. PMID 30111326